CLINICAL TRIAL: NCT03811314
Title: The Therapeutic Effect of Exercise Training on Old Patients With Dementia and Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: The Therapeutic Effect of Exercise Training on Patients With Dementia and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CF18010B
Record Dates: First submitted 2019-01-13; First posted 2019-01-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Dementia
Keywords: Dementia
MeSH Terms: conditions — Dementia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: comparison of therapeutic effect between aerobic and strength training on dementia patient, and comparison of therapeutic effect between isokinetic and isotonic training on patients with mild cognitive impairment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Strength training (Experimental): Muscle strength training programs
  Interventions: Device: Strength training
- Aerobic training (Experimental): Aerobic training programs
  Interventions: Device: Aerobic training
- Isokinetic training (Experimental): Isokinetic training
  Interventions: Device: Isokinetic trinaing
- Isotonic training (Experimental): Isotonic training
  Interventions: Device: Isotonic training

INTERVENTIONS:
Device: Strength training — Using dumbbells, butterfly machine and vertical leg press machine for strength training, 12 repetition maximum weight for 12 repetition, three times a day, five days a week, for a total of four weeks
  Arms: Strength training
Device: Aerobic training — Using stationary bicycle to perform cardiopulmonary endurance training in 50-70 heart rate reserve for 20 minutes, five days per week, for a total of four weeks
  Arms: Aerobic training
Device: Isokinetic trinaing — Using Biodex isokinetic dynanometer and set it in isokinetic mode in 60 degree per second
  Arms: Isokinetic training
Device: Isotonic training — Using Biodex isokinetic dynanometer and set it in isotonic mode at 60% of the maximal peak torque
  Arms: Isotonic training

SUMMARY:
This study aimed to clarify whether strength training or aerobic training could bring more benefits for patients with dementia, another study is to clarify whether isokinetic or isotonic training could bring more benefits for patients with mild cognitive impairment

DETAILED DESCRIPTION:
Exercise training has been evidenced to bring various of benefits for patients with dementia in past studies. However, whether strength training or aerobic training could bring better benefits has not been confirmed in the past. This study designed to recruit 30 patients with mild dementia in the first year. Every patient will receive strength training using dumbbells, butterfly machine and vertical leg press machine for four weeks. Outcome measures including self care ability, cognitive function, MCP-1, BDNF and IGF-1 levels, and the degree of depression will be recorded before and after the training. In the second year, the investigators also designed to recruit 31 patients with mild dementia. These participants will instead receive aerobic training using stationary bicycle for four weeks. The same outcome measures will be tested as in the first year. The other part of the study recruited 46 patients with mild cognitive impairment, who were randomized into either a four-week isokinetic or isotonic training program. All cases were evaluated by isokinetic peak torque, 36-item Short Form Survey (SF-36), Mini-Mental State Examination (MMSE), Barthel Index, geriatric depression scale (GDS-15), and Timed Up and Go test (TUG test) before and after each kind of training.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged above 65 years old
2. Patients with mild dementia with Mini-mental state examination scoring 15 to 26
3. Another arm is patients with mild cognitive impairment and Mini-mental state examination scoring 23 to 27

Exclusion criteria:

1. Cardiopulmonary diseases or orthopedical conditions that prohibit the patient from receiving exercise training of our programs
2. Cognitive problems that impede the patient to understand and answer the content of our questionnaires.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Barthel index | 4 weeks
  To evaluate function of activities of daily living, range from 0-100, higher values represent a better outcome
Mini-mental state examination | 4 weeks
  To evaluate cognitive function, range from 0-30, higher values represent a better outcome
Montreal Cognitive Assessment | 4 weeks
  To evaluate cognitive function, range from 0-30, higher values represent a better outcome
Geriatric Depression Scale | 4 weeks
  To evaluate patient's depression status, range from 0-15, higher values represent a worse outcome
Timed up and go test | 4 weeks
  Measure the time taken by a patient to stand up from a chair, walk three meters, return, and sit back on the chair
SF-36 | 4 weeks
  consists of 36 questions categorized into 8 subdomains, including physical functioning, role limitations due to physical health, pain, general health condition, vitality, social functioning, role limitations due to emotional problems, and emotional well-being.

SECONDARY OUTCOMES:
Concentration of serum brain derived neurotrophic factor (BDNF) | 4 weeks
  Increasing BDNF level is related to preventing neurodegeneration.
Concentration of plasma insulin-like growth factor-1 (IGF-1) | 4 weeks
  Lower plasma level of IGF-1 is associated with an increased risk of developing Alzheimer's dementia, and higher levels of it may protect against neurodegeneration.
Concentration of plasmamonocyte chemotactic protein-1 (MCP-1) | 4 weeks
  The elevation of MCP-1 concentration usually means the progression of systemic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Yang Cheng, MDPHD, Principal Investigator — Department of rehabilitation of Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Liu IT, Lee WJ, Lin SY, Chang ST, Kao CL, Cheng YY. Therapeutic Effects of Exercise Training on Elderly Patients With Dementia: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 May;101(5):762-769. doi: 10.1016/j.apmr.2020.01.012. Epub 2020 Feb 19. PMID 32084347